CLINICAL TRIAL: NCT00032656
Title: Adolescents' Use of Complementary and Alternative Medicine
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Other Study IDs: R21AT000407-01 (NIH)
Record Dates: First submitted 2002-03-27; First posted 2002-03-28 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Healthy
Keywords: Adolescents; Alternative and complimentary medication use; Health services utilization; Communication; Quality of care
MeSH Terms: conditions — Patient Acceptance of Health Care; Communication

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
The purpose of this study is to help improve our understanding of when and why adolescents decide to use alternative and complimentary medicines, and to understand factors that lead to better communication between youth and their clinicians.

DETAILED DESCRIPTION:
Alternative therapies and herbal remedies are increasingly recognized as having therapeutic value, and as many as 42% adults use some form of complementary and alternative medicine (CAM). The prevalence of CAM use among adolescents is not known. Questions remain about the safety and efficacy of some CAM therapies, and how to best facilitate communication about alternative medicine between patients and clinicians. Research with adults shows that most do not reveal their use of alternative therapies to their providers. Adolescence is a time of experimentation and the beginning of a shift from depending upon parents to taking responsibility for one's own care. Thus, the health practices begun in adolescence have an impact into adulthood. However, none of the current guidelines for the provision of care to adolescents advise asking about complementary or alternative medicine use. Finally, adolescents are exposed to increasing coverage of CAM in the media, and on the internet. The specific aims of this study are to: 1) determine the prevalence of complementary and alternative medicine use among a representative sample of adolescents, 2) describe the range of therapies adolescents use, and where they are procured, 3) describe adolescent and clinician factors that are associated with communication between adolescents and their providers about complementary and alternative medicine, and 4) describe adolescents' exposure to information about CAM from sources such as parents, providers, and the media, and how this impacts CAM use. We propose a cross sectional random digit dial telephone survey of 1200 adolescents in Monroe County, NY. Our findings will allow us to understand how adolescents use alternative medicine. Additionally, since alternative therapies can have potentially serious side-effects or drug interactions, insight into how and when alternative medicine use is disclosed may help clinicians provide better care to adolescents.

ELIGIBILITY:
Adolescents ages 14-19

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1400
Dates: Start 2001-02; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D. Klein, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Department of Pediatrics, Rochester, New York, United States